CLINICAL TRIAL: NCT02439671
Title: A Service Delivery Model to Better Support Young Adults With Autism Spectrum Disorders in the Transition From School to the Community
Brief Title: Transition Support Program for Young Adults With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Aparna Nadig, Ph.D., McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Max Bell / McGill x-209094
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Transition Support Program for young adults
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate intervention (Experimental): Participant assigned to McGill Transition Support Program in next available session
  Interventions: Behavioral: McGill Transition Support Program
- Waiting List control (No Intervention): Participant assigned to waiting list for one session prior to receiving McGill Transition Support Program in following session

INTERVENTIONS:
Behavioral: McGill Transition Support Program — The McGill Transition Support Program is manual-based, including 15 modules of curriculum, five in each of the following domains of skills:
  * Social communication (e.g. listening, perspective taking)
  * Self-determination (e.g. problem-solving, self-advocacy)
  * Working with others (e.g. knowing your context, teamwork)
  Nine out of the 15 modules are selected for each group according to the common needs endorsed by participants on a needs assessment questionnaire. Each group consists of 4 adults and two facilitators who were graduate students in Speech Language Pathology or Educational Psychology.
  The intervention follows a Self-Determination Learning Model of Instruction (SDLMI) that considers the individual's strengths and needs in the development of personal goals and plans for one's future. A workbook is used to accompany each module with the aim of having the participants practice and generalize the main content messages.
  Arms: Immediate intervention

SUMMARY:
This study investigates a service delivery model to better support young adults with autism spectrum disorders (ASD) in the transition from school to the community. The effectiveness of the "McGill Transition Support Program", a small-group format intervention (meeting once a week for 2 hours over 10 weeks) focusing on communication, self-determination and working with others skills, is measured by multiple pre- and post-program-assessments in a "staggered enrollment trial", a variant of a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The difficulties characterizing Autism Spectrum Disorder (ASD) are often associated with childhood; however, ASD is a lifespan diagnosis that continues to impact opportunities in the community. There is currently a very significant gap in support services for young adults with ASDs that has grave consequences both for individuals and their families in terms of vocational success and social inclusion and for society as a whole in terms of the financial burden of long-term adult care.

Individuals on the higher end of the autism spectrum do not have intellectual disability and possess good language skills. Yet they often show significant difficulty with applying their skills during demanding social interactions, which is detrimental to their ability to form relationships and navigate interactions in the workplace. In the few studies of outcomes of adults with ASD it is reported that fewer than 5% of adults at the highest end of the spectrum were living independently and only 12% were employed viably. This underscores the tremendous need for targeted services for young adults with ASD without intellectual disability.

The McGill Transition Support Program was developed to target participants' self-expressed needs in communication, self-determination and working with others skills, which have been associated with better quality of life. Besides the intake, pre- and post-program measures sessions, the participants, aged 18 - 30 years, take part in ten 2-hour group meetings. The study design has been termed a "staggered enrollment trial", that is participants were randomly assigned to take part in the program in the next available cycle or to the waiting list for a subsequent cycle. Pre- and post-program assessment include social problem solving stories, quality of life and self-determination measures, a communication task and a needs and skills questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* proficient and able to communicate in English
* between the ages of 18 and 30 years upon entering the study
* ASD classification according to scores on either or both the Social Communication Questionnaire-Lifetime (SCQ) and the Autism Diagnostic Observation Schedule-2 (ADOS-2, Module 4 revised algorithm)
* Either or both non-verbal IQ, assessed by Raven's Progressive Matrices, or verbal IQ assessed by Wechsler Abbreviated Scales of Intelligence, verbal subtests, in the normal range

Exclusion Criteria:

* current enrollment in another similar transition support service, that is, a group-format service that has the goals of improving the areas of social interaction and communication, self-determination and advocacy, and working with others skills

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Social problem-solving task (Channon & Crawford, 2010) | 4-6 weeks prior to session, 4-6 weeks after session
Change in Arc's Self-Determination Scale (SDS; Wehmeyer & Kelchner, 1995) | 4-6 weeks prior to session, 4-6 weeks after session, and 12 month follow-up post-Program
Change in Quality of Life Questionnaire (Shalock & Keith, 1993) | 4-6 weeks prior to session, abridged version: 4-6 weeks after session and 12 month follow-up post-Program

SECONDARY OUTCOMES:
Curriculum-specific workbook questions | every week for 9 weeks at the end of group intervention meetings
Participant Program Evaluation Survey (Flanagan & Nadig, 2012) | 4-6 weeks after Program and 12 month follow-up post-Program
  Questionnaire composed of qualitative (open-ended) questions
Parent Program Evaluation Survey (Flanagan & Nadig, 2012) | 4-6 weeks after Program
  (Questionnaire composed of quantitative (Likert-type) and qualitative (open-ended) questions)
Questionnaire on vocational, educational and living situation outcomes | 12 month follow-up post-Program
Communication task (Nadig, Vivanti, & Ozonoff, 2009) | 4-6 weeks prior to session, 4-6 weeks after session

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Nadig, Ph.D., Principal Investigator — School of Communication Sciences and Disorders, McGill University; Tara Flanagan, Ph.D., Principal Investigator — Department of Educational and Counselling Psychology, McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Background] Channon S, Crawford S. Mentalising and social problem-solving after brain injury. Neuropsychol Rehabil. 2010 Oct;20(5):739-59. doi: 10.1080/09602011003794583. Epub 2010 Jun 1. PMID 20526955
- [Background] Ganz ML. The lifetime distribution of the incremental societal costs of autism. Arch Pediatr Adolesc Med. 2007 Apr;161(4):343-9. doi: 10.1001/archpedi.161.4.343. PMID 17404130
- [Background] Mercer SL, DeVinney BJ, Fine LJ, Green LW, Dougherty D. Study designs for effectiveness and translation research :identifying trade-offs. Am J Prev Med. 2007 Aug;33(2):139-154. doi: 10.1016/j.amepre.2007.04.005. PMID 17673103
- [Background] Nadig A, Vivanti G, Ozonoff S. Adaptation of object descriptions to a partner under increasing communicative demands: a comparison of children with and without autism. Autism Res. 2009 Dec;2(6):334-47. doi: 10.1002/aur.102. PMID 19998354
- [Background] Taylor JL, Seltzer MM. Changes in the autism behavioral phenotype during the transition to adulthood. J Autism Dev Disord. 2010 Dec;40(12):1431-46. doi: 10.1007/s10803-010-1005-z. PMID 20361245
- [Background] Howlin P, Goode S, Hutton J, Rutter M. Adult outcome for children with autism. J Child Psychol Psychiatry. 2004 Feb;45(2):212-29. doi: 10.1111/j.1469-7610.2004.00215.x. PMID 14982237
- [Background] Barnard J, Harvey V, Potter D, Prior A. Ignored or ineligible? The reality for adults with autism spectrum disorders. The National Autistic Society report for Autism Awareness Week. 2001. London: NAS publications.
- [Background] Flangan T, Nadig A. Transition Support Needs Assessment. 2012
- [Background] Graetz JE. Autism grows up: opportunities for adults with autism. Disability and Society. 2010;25(1):33-47.
- [Background] Hendricks DR, Wehman P. Transition from school to adulthood for youth with autism spectrum disorders. Focus on Autism and Other Developmental Disabilities. 2009;24(2):77-88.
- [Background] Levy A, Perry A. Outcomes in adolescents and adults with autism: A review of the literature. Research in Autism Spectrum Disorders. 2011;5(4):1271-1282.
- [Background] Lord C, Rutter M, DiLavore PC, Risi S. Autism Diagnostic Observation Schedule (ADOS). 1999. Los Angeles, CA: Western Psychological Association.
- [Background] Raven J, Raven JC, Court JH. Manual for Raven's Progressive Matrices and Vocabulary Scales. 2003, updated 2004. San Antonio, TX: Pearson Assessment.
- [Background] Rutter M, Bailey A, Berument SK, Lord C, Pickles A. Social Communication Questionnaire (SCQ). 2003. Los Angeles, CA: Western Psychological Services.
- [Background] Schalock R, Keith K. Quality of Life Questionnaire. 1993, 2004 Revision. Worthington, OH: IDS Publishing.
- [Background] Wechsler D. Wechsler Abbreviated Scales of Intelligence (WASI). 1999. San Antonio, TX: The Psychological Corporation/Harcourt Assessment.
- [Background] Wehmeyer ML, Field S. Self-determination: Instructional and assessment strategies. 2007. Thousand Oaks, CA: Corwin Press.
- [Background] Wehmeyer ML. Student self-report measure of self- determination for students with cognitive disabilities. Education and Training in Mental Retardation and Developmental Disabilities. 1996;31:282-293.
- [Background] Wehmeyer ML, Kelchner K. The Arc's Self-Determination Scale. 1995. Arlington, TX: Arc National Headquarters.
- [Derived] Nadig A, Flanagan T, White K, Bhatnagar S. Results of a RCT on a Transition Support Program for Adults with ASD: Effects on Self-Determination and Quality of Life. Autism Res. 2018 Dec;11(12):1712-1728. doi: 10.1002/aur.2027. Epub 2018 Nov 19. PMID 30451392